CLINICAL TRIAL: NCT05136898
Title: A Phase 3b, Open-Label, Single-Arm, Multicenter Study to Assess the Feasibility of Home Instillation of UGN-102 for Treatment of Patients With Low-Grade (LG) Non-Muscle Invasive Bladder Cancer (NMIBC) at Intermediate-Risk (IR) of Recurrence
Brief Title: Feasibility of Home Instillation of UGN-102 for Treatment of Low-Grade (LG) Non-Muscle Invasive Bladder Cancer (NMIBC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL010
Record Dates: First submitted 2021-09-23; First posted 2021-11-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Urothelial Carcinoma Bladder
Keywords: Non-muscle invasive bladder cancer; Low grade non-muscle invasive bladder cancer; Intermediate risk non-muscle invasive bladder cancer; NMIBC; UGN-102; Mitomycin
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UGN-102 (Experimental): Patients will receive 6 once-weekly intravesical instillations of UGN-102 (75 mg mitomycin). Treatment Visit 1 will occur at the investigative site and instillation will be performed by a qualified physician. Treatment Visits 2 to 6 will occur at the patient's home and instillation will be performed by a properly trained and qualified home health professional.
  Interventions: Drug: UGN-102

INTERVENTIONS:
Drug: UGN-102 — UGN-102 consists of mitomycin and sterile hydrogel (a proprietary thermally responsive gel) that is used to reconstitute mitomycin before instillation. The reverse thermal properties of UGN-102 allow for local administration of mitomycin as a liquid under chilled conditions, with subsequent conversion to a semi-solid gel depot following instillation into the bladder.
  Other Names: UGN-102 (mitomycin) for intravesical solution

SUMMARY:
This study aims to demonstrate that home instillation of UGN-102 is a feasible alternative to instillation in a clinical setting, which might mitigate patient challenges (logistical, expense, and comfort) when receiving treatment for low-grade intermediate-risk non-muscle invasive bladder cancer (LG-IR-NMIBC).

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the feasibility of home instillation of UGN-102 as an alternative to instillation in a clinical setting. Feasibility was assessed by evaluation of safety and tolerability, rate of discontinuation from at home study treatment, and feedback from patients, home health professionals (HHPs), and investigators via standardized questionnaires. The secondary objective of this study was to evaluate the efficacy of UGN-102 for treatment of LG-IR-NMIBC following home instillation. Efficacy was assessed at the 3-month Visit (3 months after the first instillation of UGN-102) by the complete response rate (CRR), defined as the proportion of patients who achieved a complete response (CR) as determined by cystoscopy, for cause biopsy, and urine cytology.

Patients who provided informed consent underwent a Screening Visit to determine eligibility. Screening procedures were to provide evidence of LG-NMIBC and to rule out evidence of high-grade (HG) disease.

Eligible patients were to receive 6 once-weekly intravesical instillations of UGN-102. The first instillation was performed at the investigative site and subsequent instillations were performed at the patient's home by a trained HHP. The HHP was to call the patient 1 to 2 days after each home instillation of UGN-102 to monitor for safety.

At each home instillation visit, the patient and HHP were to complete a feasibility questionnaire. In addition, the patient and investigator were to complete a feasibility questionnaire at the 3-month Visit (end of study) or Early Termination Visit.

Patients were to return to the clinic for the 3-month Visit for determination of response to treatment. Response was determined based on visual evaluation by cystoscopy (white light) (appearance, number, and size of any remaining lesions), interpretation of urine cytology, and for cause biopsy and histopathology of any remaining lesions. Any lesions or suspect tissue were to be biopsied to evaluate for persistence of disease.

Safety was evaluated based on review of adverse events (AEs), laboratory assessments, vital signs, and physical examination.

A patient was considered to have completed the study if the patient completed the 3-month Visit. Following the 3-month Visit, all patients exited the study and continued with standard of care according to their treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and the protocol.
2. Patient who has newly diagnosed or historic LG-NMIBC (Ta) histologically confirmed by cold cup biopsy at Screening or within 8 weeks before Screening.
3. Has IR disease, defined as having 1 or 2 of the following:

   * Presence of multiple tumors.
   * Solitary tumor > 3 cm.
   * Recurrence (≥ 1 occurrence of LG-NMIBC within 1 year of the current diagnosis at the initial Screening Visit).
4. Negative voiding cytology for HG disease within 6 weeks before Screening.
5. Has adequate organ and bone marrow function as determined by routine laboratory tests:

   * Leukocytes ≥ 3,000/μL (≥ 3 × 10^9/L).
   * Absolute neutrophil count ≥ 1,500/μL (≥ 1.5 × 10^9/L).
   * Platelets ≥ 100,000/μL (≥ 100 × 10^9/L).
   * Hemoglobin ≥ 9.0 g/dL.
   * Total bilirubin ≤ 1.5 × ULN.
   * AST and ALT ≤ 2.5 × ULN.
   * Alkaline phosphatase ≤ 2.5 × ULN.
   * Estimated glomerular filtration rate ≥ 30 mL/min.
6. Has no evidence of active urinary tract infection at the Screening and baseline visits.
7. Patient is willing to receive instillations of UGN-102 at home (ie, Treatment Visits 2 to 6) by an appropriately trained home health professional.
8. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for clinical study participants. Women of childbearing potential (defined as premenopausal women who have not been sterilized), including female patients and female partners of male patients, must be willing to use 2 acceptable forms of effective contraception from first instillation through 6 months post treatment. Acceptable methods of birth control that are considered to have a low failure rate (ie, less than 1% per year) when used consistently and correctly include implants, injections, combined (estrogen/progesterone) oral contraceptives, intrauterine devices (only hormonal), condoms with spermicide, sexual abstinence, or vasectomized partner.
9. Has an anticipated life expectancy of at least the duration of the trial.

Exclusion Criteria:

1. Received Bacillus Calmette-Guérin treatment for urothelial carcinoma (UC) within previous 1 year.
2. History of HG bladder cancer (papillary or carcinoma in situ) in the past 2 years.
3. Known allergy or sensitivity to mitomycin that in the investigator's opinion cannot be readily managed.
4. Clinically significant urethral stricture that would preclude passage of a urethral catheter.
5. History of:

   * Neurogenic bladder.
   * Active urinary retention.
   * Any other condition that would prohibit normal voiding.
6. Past or current T1 UC, muscle invasive UC (ie, T2, T3, T4), metastatic UC, or concurrent upper tract UC.
7. Has an underlying substance abuse or psychiatric disorder such that, in the opinion of the investigator, the patient would be unable to comply with the protocol.
8. History of prior treatment with an intravesical chemotherapeutic agent in the past 2 years except for a single dose of chemotherapy immediately after any previous TURBT.
9. Has participated in a study with an investigational agent or device within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Raju, MBBS, Study Director — UroGen Pharma
Locations (5):
- United States (5):
  - Urology Centers of Alabama (UCA), Homewood, Alabama
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Medication Management, Greensboro, North Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Virginia Urology, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- UGN-102: 6 once-weekly intravesical instillations of UGN-102 (75 mg mitomycin).
Period: Overall Study
Arm/Group | UGN-102
Started | 8
Completed | 6
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: All patients who received any dose of UGN-102.
Arm/Group | UGN-102
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 75 [55 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Previous Low-grade (LG) Non-muscle Invasive Bladder Cancer (NMIBC) Episode(s) [Count of Participants; unit: Participants]
  Yes | 8
  No | 0
Previous LG-NMIBC Episode(s) Within 1 Year [Count of Participants; unit: Participants]
  Yes | 6
  No | 2
Prior Transurethral Resection of Bladder Tumor (TURBT) [Count of Participants; unit: Participants]
  Yes | 8
  No | 0
Tumor Burden [Count of Participants; unit: Participants]
  ≤ 3 cm | 4
  > 3 cm | 4
Tumor Count [Count of Participants; unit: Participants]
  Single | 3
  Multiple | 5
Smoking History [Count of Participants; unit: Participants]
  Yes | 5
  No | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation, and TEAEs of Special Interest.
Description: The number of patients with each type of event will be summarized. TEAEs were defined as adverse events (AEs) that occurred on or after the day of the first instillation of UGN-102 or pre-treatment AEs that worsened during the study.
Time Frame: Up to 3 months
Population: All patients who received any dose of UGN-102.
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 8
Participants
  Any TEAEs | 8
  Any serious TEAEs | 3
  Any TEAEs leading to discontinuation | 2
  Any TEAEs of special interest | 7

2. Primary Outcome: Number of Participants With Post-baseline Potentially Clinically Significant (PCS) Laboratory Values
Description: PCS laboratory criteria were defined for the following parameters:
  Hematology
  * Hemoglobin < 0.8 × lower limit of normal and > 20% decrease from baseline or > 1.3 × upper limit of normal (ULN) and > 30% increase from baseline.
  * Leukocytes ≤ 2.8 or ≥ 16 × 10^3/µL.
  * Lymphocytes < 0.5 or > 20 × 10^3/µL.
  * Neutrophils < 1.0 × 10^3/µL.
  * Platelets < 75 or ≥ 700 × 10^3/µL.
  Chemistry
  * Creatinine > 2.2 mg/dL.
  * Sodium ≤ 130 or > 150 mEq/L.
  * Potassium < 3.0 or > 5.5 mEq/L.
  * Total bilirubin > 1.5 × ULN.
  * Alanine aminotransferase (ALT) > 3 × ULN.
  * Aspartate aminotransferase (AST) > 3 × ULN.
  * Gamma glutamyl transferase > 2.5 × ULN.
Time Frame: Up to 3 months
Population: All patients who received any dose of UGN-102 and who had a post-baseline laboratory value.
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 8
Participants
  Hematology | 0
  Chemistry | 0

3. Primary Outcome: Composite Score for the Post-instillation Patient Questionnaire
Description: Patients were asked to rate their experience receiving UGN-102 at home after each instillation was completed. A total of 5 domains (8 questions) were assessed:
  * Comfort (3 questions, possible range from 3 "least favorable" to 12 "most favorable").
  * Safety/concerns (1 question, possible range from 1 "least favorable" to 4 "most favorable").
  * Communication (2 questions, possible range from 2 "least favorable" to 8 "most favorable").
  * Preference compared to office instillation (1 question, possible range from 1 "least favorable" to 4 "most favorable").
  * Overall experience/satisfaction (1 question, possible range from 1 "least favorable" to 4 "most favorable").
  A composite score (sum of all 8 question scores) was also calculated (possible range from 8 "least favorable" to 32 "most favorable").
Time Frame: Up to 5 weeks
Population: All patients who received any dose of UGN-102.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | UGN-102
Number analyzed (Participants) | 8
score on a scale
  Post 2nd instillation | 32 [26 to 32]
  Post 3rd instillation: number analyzed (Participants) | 7
  Post 3rd instillation | 32 [30 to 32]
  Post 4th instillation | 32 [30 to 32]
  Post 5th instillation: number analyzed (Participants) | 6
  Post 5th instillation | 32 [30 to 32]
  Post 6th instillation: number analyzed (Participants) | 6
  Post 6th instillation | 32 [29 to 32]

4. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of patients who achieved a complete response (CR) at the 3-month Visit. A patient was considered a CR if there was no detectable disease in the bladder based on visual observation (white light cystoscopy), biopsy of remaining lesions, if applicable, and voiding urine cytology.
Time Frame: 3 months
Population: All patients who received any dose of UGN-102.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UGN-102
Number analyzed (Participants) | 8
percentage of participants | 75.0 [34.9 to 96.8]

5. Primary Outcome: Responses to the Post-instillation Home Health Professional Questionnaire
Description: Home health professionals (HHPs) were asked to share their experience administering UGN-102 at the patient's home after each instillation was completed. A total of 4 domains (4 questions) were assessed:
  * Comfort - Were you comfortable performing the instillation at this patient's home, yes (most favorable) or no (least favorable)?
  * Difficulty - Was it difficult to perform the instillation at this patient's home, yes (least favorable) or no (most favorable)?
  * Safety/concerns - Did you have any concerns performing the instillation in the home setting, yes (least favorable) or no (most favorable)?
  * Adequate support - Did you have sufficient support performing the instillation in the home setting, yes (most favorable) or no (least favorable)?
  The number of patients whose HHP had a "most favorable" response to all 4 questions is summarized for each home instillation.
Time Frame: Up to 5 weeks
Population: All patients who received any dose of UGN-102.
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 8
Participants
  Post 2nd instillation | 8
  Post 3rd instillation | 7
  Post 4th instillation | 7
  Post 5th instillation: number analyzed (Participants) | 7
  Post 5th instillation | 7
  Post 6th instillation: number analyzed (Participants) | 6
  Post 6th instillation | 5

6. Primary Outcome: Responses to End of Study Patient and Investigator Questionnaires
Description: Patient recommendations regarding home instillation of UGN-102 were collected at the 3-month Visit or Early Termination Visit. Two questions were asked:
  * Will you recommend home instillations of UGN-102 for other patients with NMIBC, yes (most favorable) or no (least favorable)?
  * Will you recommend home instillations of UGN-102 instead of having transurethral resection of bladder tumor (TURBT) for other patients with NMIBC, yes (most favorable) or no (least favorable)?
  The number of patients who had a "most favorable" response is summarized by question.
  In addition, investigators were asked if the experience of having their patient receive instillations at home was less difficult (most favorable), more difficult (least favorable), or not different than having them receive instillations in the office. All responses are summarized.
Time Frame: 3 months
Population: All patients who received any dose of UGN-102 and who completed the end of study questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 6
Participants
  Recommend home instillations of UGN-102 for other NMIBC patients = yes | 5
  Recommend home instillations of UGN-102 instead of having TURBT = yes | 5
  Having patient receive instillations at home is less difficult than in office | 0
  Having patient receive instillations at home is more difficult than in office | 1
  Having patient receive instillations at home is not different than in office | 5

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: Per protocol, sites were instructed to report AEs that occurred from the time of informed consent to the 3-month Visit.
Arm/Group | UGN-102
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UGN-102 (N=8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UGN-102 (N=8)
Dysuria (Renal and urinary disorders) | 2
Fatigue (General disorders) | 2
Hypertonic bladder (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Anxiety (Psychiatric disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Pneumonia (Infections and infestations) | 1
Pollakiuria (Renal and urinary disorders) | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Urine flow decreased (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT05136898/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT05136898/SAP_001.pdf